CLINICAL TRIAL: NCT04505085
Title: Active Dads Healthy Families: Promoting Physical Activity and Enhancing Father-child Relationships Through Parks and Recreation
Brief Title: Active Dads Healthy Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00106052
Record Dates: First submitted 2020-07-30; First posted 2020-08-07 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Health Behavior
Keywords: physical activity; parenting; exercise; family-based; father
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: A non-randomized quasi-experimental design will be used to evaluate the feasibility of the Active Dads Healthy Families intervention, and provide preliminary data of changes over time and between two forms of the intervention. The investigators will recruit two cohorts totaling 30 father-child dyads (15 per cohort) to take part in the 8-week program delivered by Parks and Recreation. The primary outcome is program feasibility.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Dads Healthy Families: Outdoor Education (Experimental): The intervention will include outdoor education and physical activity opportunities at various outdoor parks. The program will be held one day a week for eight consecutive weeks. Parks and Recreation will facilitate and run the program. Each session will last 60 minutes and include a brief educational discussion and opportunities for various games and activities. Each session will have a special theme relevant to the outdoors. Families will also receive a home toolbox to facilitate activity and learning outside of the program. Feedback on physical activity will be provided at the beginning and the end of the program.
  Interventions: Behavioral: Active Dads Healthy Families: Outdoor Education
- Active Dads Healthy Families: Fitness (Experimental): The intervention will include physical activity opportunities at a community center. The program will be held one day a week for eight consecutive weeks. Parks and Recreation will facilitate and run the program. Each session will last 60 minutes and include a brief educational discussion and opportunities for various games and activities. Families will also receive a home toolbox to facilitate activity outside of the program. Feedback on physical activity will be provided at the beginning and the end of the program.
  Interventions: Behavioral: Active Dads Healthy Families: Fitness

INTERVENTIONS:
Behavioral: Active Dads Healthy Families: Outdoor Education — The intervention will include outdoor education and physical activity opportunities at various outdoor parks. The program will be held one day a week for eight consecutive weeks. Parks and Recreation will facilitate and run the program. Each session will last 60 minutes and include a brief educational discussion and opportunities for various games and activities. Each session will have a special theme relevant to the outdoors. Families will also receive a home toolbox to facilitate activity and learning outside of the program. Feedback on physical activity will be provided at the beginning and the end of the program.
  Arms: Active Dads Healthy Families: Outdoor Education
Behavioral: Active Dads Healthy Families: Fitness — The intervention will include physical activity opportunities at a community center. The program will be held one day a week for eight consecutive weeks. Parks and Recreation will facilitate and run the program. Each session will last 60 minutes and include a brief educational discussion and opportunities for various games and activities. Families will also receive a home toolbox to facilitate activity outside of the program. Feedback on physical activity will be provided at the beginning and the end of the program.
  Arms: Active Dads Healthy Families: Fitness

SUMMARY:
The purpose of this study is to evaluate the feasibility of implementing a community-delivered physical activity program for fathers and their children ages 2-5 years.

DETAILED DESCRIPTION:
The investigators will evaluate the feasibility of a community-based father-child physical activity promotion program. The investigators will work with a local Parks and Recreation department to recruit and deliver programming to three cohorts of fathers and their children 2-5 years old. To evaluate program feasibility, the investigators will assess recruitment efforts, program attendance, and participant engagement and satisfaction with the program. The investigators will also assess change in father-child outcomes post program including objectively measured physical activity, fathers' parenting, and father involvement.

ELIGIBILITY:
Inclusion Criteria:

* Father or father figure to child between the ages 2-5 years
* Father or father figure 18+ years
* Can speak and read in English

Exclusion Criteria:

* Father or child has a physical disability precluding them from being physically active

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-17 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Recruitment as measured by number of participants who enroll | Baseline
Attendance as measured by number of participants present at each session | Baseline through 8 weeks
Degree of participation in physical activity during each session | Baseline through 8 weeks
  As measured by observation using the System for Observing Fitness Instruction Time (SOFIT) instrument, activity scores range from 1 "lying down" to 5 "vigorous"
Percent of participants satisfied with the program as measured by self-report evaluation survey | 8 weeks
  Self-report program evaluation survey; 13 items with responses ranging from 1 "strongly disagree" to 5 "strongly agree"
Percent of participants who complete all study measures | Baseline
Percent of participants who complete all study measures | 8 weeks

SECONDARY OUTCOMES:
Change in moderate to vigorous physical activity as measured by accelerometry | Baseline, 8 weeks
  Child objectively measured physical activity
Change in moderate to vigorous physical activity as measured by accelerometry | Baseline, 8 weeks
  Father objectively measured physical activity
Change in father support for child physical activity as measured by father self-report | Baseline, 8 weeks
  15-item engagement subscale score from the Preschool Physical Activity Parenting Practices instrument, scored by calculating mean of items (range 1-5), higher scores indicate greater parent engagement
Change in father physical activity psychological control as measured by father self-report | Baseline, 8 weeks
  5-item psychological control subscale score from the Preschool Physical Activity Parenting Practices instrument, scored by calculating mean of items (range 1-5), higher scores indicate greater parent psychological control
Change in father involvement in physical play as measured by father self-report | Baseline, 8 weeks
  9-item scale about father involvement in physical play, scored by calculating the mean of all items (range 1-6), with higher scores indicating greater father involvement
Change in father involvement in care-giving as measured by father self-report | Baseline, 8 weeks
  13-item scale about father involvement in care-giving, scored by calculating the mean of all items (range 1-6), with higher scores indicate greater father involvement

CONTACTS AND LOCATIONS:
Overall Officials: Sarah C Armstrong, MD, Principal Investigator — Duke University
Locations (1):
- Durham Parks and Recreation, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No